CLINICAL TRIAL: NCT00889278
Title: Higher Infused Lymphocyte Counts Improve Antibody Response to Immunization After Autologous Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Richard Zuckerman, Director, Transplant Infectious Disease Program, Dartmouth-Hitchcock Medical Center
Other Study IDs: D0748
Record Dates: First submitted 2009-04-24; First posted 2009-04-28 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Lymphoma
Keywords: Lymphoma; Autologous Peripheral Blood Stem Cell Transplant; APBSCT; Pneumococcal Conjugate Vaccine
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 10cc Peripheral Blood
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine if higher absolute lymphocyte count in the infused stem cell autograft (A-ALC) will lead to an improved antibody response to post-transplant immunization with Pneumococcal Conjugate Vaccine and permit effective immunization at 6 months post-transplant in lymphoma patients receiving Autologous Peripheral Blood Stem Cell Transplantation.

DETAILED DESCRIPTION:
Infectious diseases remain a leading cause of morbidity and mortality in patients who receive high-dose chemotherapy followed by Autologous Peripheral Blood Stem Cell Transplantation (APBSCT). Infectious disease complications of transplantation might be reduced by effective post-transplant immunization but reconstitution of the immune system may take months to years after transplantation and responses to immunization are often attenuated in this setting. Correlates of improved immune reconstitution and response to immunization after transplantation would be important to identify. It has been recently shown that higher absolute lymphocyte count in the infused stem cell autograft (A-ALC) and higher ALC at day +15 after stem cell infusion (ALC-15) are independently associated with improved overall survival after APBSCT. The mechanism of this association is unclear, but this finding suggests that improved immune responses to immunization might also be achieved with this approach making it possible to immunize at 6 months instead of at one year. This hypothesis has never been evaluated.

Survival following APBSCT is improved with a higher A-ALC and ALC-15. It is postulated that the higher lymphocyte numbers correlate with improved immune surveillance and destruction of minimal residual disease. Thus, one must consider the probability higher A-ALC will confer improved response to T-cell dependent immunization early after transplant.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Lymphoma or lymphoproliferative disease diagnosis
* Scheduled APBSCT
* Able to give informed consent and comply with the procedures of the study
* Enrollment in other interventional trials are allowed at the discretion of the investigators

Exclusion Criteria:

* Contraindication to Prevnar®
* Has received immune globulin within 5 months prior to being enrolled on the study or plans to receive immune globulin prior to the day +270 (+/-30) visit
* Currently participating in, or scheduled to participate in any clinical trial using investigational immune modulators (e.g. IL-2) at any time prior to the completion of follow-up in this study.
* Any other underlying medical condition that, in the opinion of the investigator, may interfere with the evaluation of study objectives
* Day +180(+/- 30days) Eligibility:
* Has received immune globulin within the past 5 months prior to the receipt of the vaccine or plans to receive immune globulin prior to the day +270(+/- 30) visit
* Is pregnant (as determined by urine or serum B-HCG test)
* Participant has a contraindication to Prevnar®
* A recent (<72 hours) febrile illness (axillary temperature >99.5°F [>37.5°C], oral temperature >100.3oF [>37.9oC], or rectal temperature >101.3°F[>38.5°C]) prior to the study vaccination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lymphoma patients of Dartmouth Hitchcock Medical Center's Norris Cotton Cancer Center schedule to receive APBSCT.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-02 (Actual); Primary Completion 2012-03-01 (Actual); Study Completion 2016-01-05 (Actual)

PRIMARY OUTCOMES:
Antibody response to vaccination | 2 Years
  To assess the antibody response to Prevnar® and its correlation to autograft absolute lymphocyte count (A-ALC).

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Zuckerman, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States